CLINICAL TRIAL: NCT02046941
Title: Brain Biomarkers of Response to Treatment for Apraxia of Speech
Acronym: SPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C1532-I
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Aphasia; Stroke
Keywords: aphasia; stroke; Magnetic Resonance Imaging; Diffusion Magnetic Resonance Imaging
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Speech Production Treatment (Experimental): This treatment employs a response-contingent hierarchy made up of verbal modeling/repetition, graphic cueing, integral stimulation, and articulatory placement instruction. The investigators chose this treatment for the following reasons: 1) rigor of development demonstrated across multiple studies, 2) large and predictable effects with published, quantified effect sizes, 3) a demonstrated pattern of generalization to untrained items, illustrating experimental control, 4) an established multi-modal stimulation protocol, and 5) use of repeated practice, which is associated with neural plasticity.
  Interventions: Behavioral: Speech Production Treatment

INTERVENTIONS:
Behavioral: Speech Production Treatment — This treatment employs a response-contingent hierarchy made up of verbal modeling/repetition, graphic cueing, integral stimulation, and articulatory placement instruction.

SUMMARY:
The study will use MRI brain imaging to identify brain changes associated in stroke patients after they receive speech-language treatment for their speech difficulties.

DETAILED DESCRIPTION:
The goals of the current study are to identify grey and white matter regions that are predictive of speech treatment response and measure neural plasticity in response to speech treatment, using state-of-the-art neuroimaging and statistical processing techniques in a group of well-characterized left hemisphere patients meeting strict inclusionary criteria. Specifically, the investigators will use voxel-based lesion symptom mapping to identify lesion sites most predictive of a positive response to speech treatment and advanced diffusion imaging techniques to map changes in the integrity of white matter tracts from pre- to post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are age 40-90
* primary English speaker since < age 5
* a history of a single left hemisphere stroke
* at least 1 year post-stroke
* at least 12 years of education
* pre-morbidly right-handed (Edinburgh Handedness Questionnaire)
* within normal limits on the Test of Non-Verbal Intelligence

Exclusion Criteria:

* Exclusion criteria will include a pre-morbid neurologic or psychiatric history
* history/current substance abuse disorder
* MRI contraindications
* other motor speech disorders (e.g., dysarthria)
* current or recent (<2 months) speech/language therapy
* prior SPT
* pre-morbid history of speech/language disorders
* significant hearing disabilities (based on a pure-tone audiological screen at 35 dB HL at 500, 1K, and 2K Hz for at least one ear)
* aphasia severity resulting in <30th percentile performance on the Porch Index of Communicative Ability-R

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana V. Baldo, PhD, Principal Investigator — VA Northern California Health Care System, Mather, CA
Locations (1):
- VA Northern California Health Care System, Mather, CA, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Speech Production Treatment
Started | 17
Completed | 10
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Speech Production Treatment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent of Trained Items Correctly Repeated
Description: For each participant, three target sounds were chosen: single consonants, vowels, or clusters at the word level. Based on these target sounds, 10 word items were generated for each target sound that served as Trained Items. Participants were tested on lists of Trained Items (probe trials) during repeated sessions in pre-intervention stage to establish baseline performance (percent of each word list repeated correctly) and during every other treatment session (again, percent of each word list repeated correctly). The change in percent correct list repetition from pre-intervention (5 probe trials) to the end of intervention (final 3 probe trials) was calculated as individual treatment effect sizes using the Busk & Serlin (1992) d2 statistic, which involves subtracting the difference between mean performance at end of the intervention minus pre-intervention, divided by the pooled standard deviation of the two phases. The larger the d2 effect size, the larger the effect of the treatment.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: d2 treatment effect size
Arm/Group | Speech Production Treatment
Number analyzed (Participants) | 10
d2 treatment effect size | 6.67 (4.43)

2. Primary Outcome: Change From Baseline in Percent of Untrained Items Correctly Repeated
Description: To test generalization, we assessed the change in performance (percent correct repetition) on lists of 10 Untrained Items that had the same speech production targets as each patient's lists of 10 Trained Items, balanced for syllabic structure, word frequency, grammatical form class, and stress pattern. Just as for Trained Items, participants were tested on the lists of Untrained Items (probe trials) during repeated sessions in the pre-intervention stage to establish baseline performance and during every other treatment session (percent of each word list repeated correctly). The change in percent correct list repetition from pre-intervention (5 probe trials) to end of intervention (final 3 probe trials) was calculated as individual treatment effect sizes using the d2 statistic: the difference between mean performance at end of the intervention minus pre-intervention, divided by the pooled standard deviation. The larger the d2 effect size, the larger the effect of the treatment.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: d2 treatment effect size
Arm/Group | Speech Production Treatment
Number analyzed (Participants) | 10
d2 treatment effect size | 2.66 (4.39)

3. Secondary Outcome: Percentage Change in Fractional Anisotropy (FA)
Description: To measure neuroplasticity associated with the speech treatment protocol, the investigators calculated the percent change in fractional anisotropy (FA) from pre- to post-treatment for each of the eight fiber tracts in the left hemisphere. The average percentage change in FA across all eight fiber tracts was calculated, which could thus range from 0-100%. A positive change indicates an increase in white matter integrity, and a negative change indicates a decrease in white matter integrity. A number close to 0 indicates minimal/no significant change.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: average percent change in FA
Arm/Group | Speech Production Treatment
Number analyzed (Participants) | 10
average percent change in FA | -0.46 (1.05)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Same AE reporting description as clinicaltrials.gov.
Arm/Group | Speech Production Treatment
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
The generalizability of the study is limited due to the small sample size. However, published studies using this treatment intervention include even smaller samples (3-4 patients), due to the time-intensive nature of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2014-01-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT02046941/Prot_000.pdf
  • Statistical Analysis Plan (2014-01-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT02046941/SAP_001.pdf